CLINICAL TRIAL: NCT00198653
Title: Newborn Thermal Care Practices in Rural India: A Community Based Program to Prevent and Improve Recognition and Management of Hypothermia
Brief Title: Newborn Thermal Care Practices: A Community Based Program to Prevent Hypothermia
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: H.22.02.07.15.A1
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2007-05-07 (Estimated); Status verified 2007-04

CONDITIONS: Hypothermia
Keywords: Hypothermia; Newborn; India; Maternal/Child Health; Infant; Kangaroo Mother Care
MeSH Terms: conditions — Hypothermia

INTERVENTIONS:
Behavioral: Newborn Thermal Care Practice

SUMMARY:
The purpose of this study is to train mothers/caretakers on how to prevent their babies from becoming too cold.

DETAILED DESCRIPTION:
This study is designed to determine domiciliary care knowledge, attitudes and practices regarding essential newborn care, with a focus on newborn thermal control; develop behavior change communications to promote prevention, early recognition and effective management of newborn hypothermia, evaluate impact and cost-effectiveness of education/behavior change communications delivered by Community Health Workers and Community Health Promoters/Change Agents on essential newborn care practices, including care-seeking; prevalence, recognition and management of hypothermia, including adaptation, safety and utility of Kangaroo Mother Care; and neonatal morbidity and mortality; evaluate the feasibility and acceptability of using LCT ThermoSpot device in rural communities to enhance mothers' recognition and management of neonatal hypothermia; determine the influence of the neonatal hypothermia indicator (ThermoSpot) on recognition of and response to newborn hypothermia and health-seeking behavior of the caregivers; develop algorithms for recognition and management of hypothermia to inform neonatal IMCI and verbal autopsy protocols and gain insight into the potential roles of various cadres of workers in providing neonatal health services at the community level and inform the development of models of community-based essential newborn care.

ELIGIBILITY:
Inclusion Criteria:

* Uttar Pradesh
* Newborns at home

Exclusion Criteria:

* Hospitalized babies

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Dates: Start 2003-03; Study Completion 2006-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gary Darmstadt, MD, Principal Investigator — Johns Hopkins Bloomberg School of Public Health
Locations (1):
- CSMMU at Lucknow; King Georges Medical College, Lucknow, Uttar Pradesh, India

REFERENCES:
- [Derived] Kumar V, Mohanty S, Kumar A, Misra RP, Santosham M, Awasthi S, Baqui AH, Singh P, Singh V, Ahuja RC, Singh JV, Malik GK, Ahmed S, Black RE, Bhandari M, Darmstadt GL; Saksham Study Group. Effect of community-based behaviour change management on neonatal mortality in Shivgarh, Uttar Pradesh, India: a cluster-randomised controlled trial. Lancet. 2008 Sep 27;372(9644):1151-62. doi: 10.1016/S0140-6736(08)61483-X. PMID 18926277